CLINICAL TRIAL: NCT05182775
Title: A Clinical Research on the Use of Fecal Bacteria Transplantation for Treatment of IgA Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Provincial People's Hospital (Other Government)
Responsible Party: Principal Investigator, 李亚峰, Professor, Shanxi Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanxiPPH
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-11

CONDITIONS: IgA Nephropathy
Keywords: IgAN; FMT
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: Case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): This trial is a prospective study without a control group. It is planned to recruit 15 patients with IgA nephropathy. The experimental group received fecal bacteria transplantation through FMT capsule. The researchers will judge the effectiveness and safety of fecal bacteria transplantation in the treatment of IgA nephropathy by observing the changes of monitoring indicators before and after fecal bacteria transplantation and during follow-up. Donor screening and FMT capsule preparation were completed by Dongyuan Yikang company (www.dongyuanyikang. com).The patients participating in the trial took 16 Enterobacteriaceae capsules on day 1, day 8 and day 15 respectively as a course of treatment. The researchers will collect stool samples from patients one day before taking the medicine, one week after the last taking the medicine and one month after the last taking the medicine, and analyze the intestinal flora by sequencing
  Interventions: Procedure: Fecal bacteria transplantation

INTERVENTIONS:
Procedure: Fecal bacteria transplantation — Fecal microbiota transplantation (FMT) refers to the transplantation of functional flora from the feces of a healthy person into the gastrointestinal tract of a patient, thereby reestablishing the intestinal flora with normal function. FMT promotes the treatment of intestinal microecology by eliminating single microorganisms or certain pathogens (such as vaccines and antibiotics) and increasing beneficial bacteria (such as prebiotics and probiotics) to the reconstruction of intestinal microecology. The best treatment indication for FMT is Clostridium difficile infection, which is a treatment choice confirmed by expert consensus and guidelines in many countries and regions. Meanwhile, FMT has been used in the treatment and research of many intestinal microbiome related diseases worldwide.

SUMMARY:
The role and related mechanisms of gut microecology in the development and progression of IgA nephropathy were investigated by treating IgA nephropathy subjects with oral probiotic capsules (FMT) combined with metagenomic sequencing and metabolomic analysis.

DETAILED DESCRIPTION:
IgA Nephropathy (IgAN) is a serious threat to human health. The exact pathogenesis of IgAN has not been elucidated yet. Currently, there is no specific and effective treatment except supportive therapy based on renin angiotensin system inhibitor. IgAN is characterized by IgA deposits in the mesangial of the kidney, persistent hematuria, and often associated with respiratory or gastrointestinal infections. Recent studies have shown a link between human genetics, gut microbiology and the pathogenesis of IgAN. Patients with kidney disease are often accompanied by intestinal flora disorder, and intestinal flora disorder will accelerate the process of kidney disease. In recent years, multiple omics studies have found that mucosal microbial immunity is involved in the pathogenesis of IgAN, among which respiratory tract and digestive tract infections can cause or aggravate IgAN. Sporadic studies have shown that intestinal microbiome diversity in IgAN patients is lower than that in normal subjects. In IgAN patients, the abundance of beneficial bacteria such as Clostridium, Enterococcus and Lactobacillus is significantly reduced. The abundance of Ruminococcus, Lachnospiraceae and Streptococcaeae increased significantly. Previous studies by the research team confirmed a strong correlation between human genetic background, intestinal microecology, and IgAN pathogenesis. Nine Single nucleotide polymorphisms (SNPS) were associated with IgAN in 1511 IgAN patients and 4469 healthy controls. Among them, the dangerous type of genes and the intestinal bacteria (Dialister/Bacilli) reduce harmful bacteria and is associated with increased (Erysipelotrichaceae/Lachnobacterium). Using metagenomic high-throughput sequencing technology, the team further studied the intestinal microflora structure at the species level in 16 IgAN patients confirmed by biopsy and 32 healthy individuals, and showed significant differences in composition and relative abundance between the two groups. The abundance of Ruminococcus gnavus, a subgenus of Ruminococcus, increased significantly in IgAN patients. Correlation analysis showed that there was a significant positive correlation between active rumen coccus and serum IgA and pathological severity in IgAN patients. Fecal microbiota transplantation (FMT) refers to the transplantation of functional flora from the feces of a healthy person into the gastrointestinal tract of a patient, thereby reestablishing the intestinal flora with normal function. FMT promotes the treatment of intestinal microecology by eliminating single microorganisms or certain pathogens (such as vaccines and antibiotics) and increasing beneficial bacteria (such as prebiotics and beneficial bacteria) to the reconstruction of intestinal microecology. The best treatment indication for FMT is Clostridium difficile infection, which is a treatment choice confirmed by expert consensus and guidelines in many countries and regions. Meanwhile, FMT has been used in the treatment and research of many intestinal microbiome related diseases worldwide. Since the occurrence of IgAN is related to intestinal flora, we attempted to conduct fecal bacteria transplantation by using FMT capsules in patients with IgA nephropathy, so as to explore the effectiveness and safety of FMT in the treatment of IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subjects: IgA nephropathy patients diagnosed by renal biopsy (2) After 3 ~ 6 months of ACEI / ARB treatment, urinary protein was still > 0.5g/d (3) eGFR30 120ml/min/1.73 ㎡ (4) Unable to tolerate the side effects of glucocorticoids and immunosuppressants (5) If the urine pregnancy test is negative and there is no pregnancy plan in the next 18 months, effective contraceptive measures can be taken (6) Age: 18-70 years old (7) Inpatient (8) Sign the informed consent form for clinical research and the informed consent form for patients treated with flora transplantation (FMT)

Exclusion Criteria:

* (1) Secondary IgA nephropathy: such as SLE, liver cirrhosis, IgA vasculitis (2) Antibiotics in recent 14 days (3) Malignant hypertension or other uncontrollable severe hypertension (systolic blood pressure > 160mmhg or diastolic blood pressure > 110mmhg) (4) Active systemic infection or serious infection within 1 month before enrollment, including HIV, HBV and HCV (5) Leukocyte count < 3.0x109 / L, or anemia (hemoglobin < 80g / L); Platelet count < 80x10 9 / L,Or other blood system diseases (6) There were malignant tumors and other diseases, and the expected survival time was < 3 months (7) Severe cardiovascular and cerebrovascular diseases and intestinal dysfunction (8) There are other immune system diseases (9) Presence of IBD, CDI, or gastrointestinal tumors (10) There is active gastrointestinal bleeding or acute and chronic gastrointestinal inflammation (11) Being or having received FMT (12) Psychosis and cognitive impairment (13) History of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
24-hour urinary protein quantification | 6 months after the end of the trial
  Percentage of subjects with 24-hour urinary protein quantification < 0.5g/d

SECONDARY OUTCOMES:
BP | 6 months after the end of the trial
  Percentage of subjects with BP < 130 / 80mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ya-feng Li, Professor, Principal Investigator — Shanxi Medical University
Locations (1):
- Shanxi Provincial People's Hospita, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The Electronic Data Capture (EDC) system developed by national Cardiovascular Center was used to collect trial Data. EDC system has been rigorously tested and fully meets the requirements of "Quality Management Specifications for Drug Clinical Trials" and "Technical Guide for Clinical Trial Data Management". Before the system is officially launched, relevant users should be trained and tested to ensure that the system meets the test requirements. After the official launch, relevant personnel will be given the account and password. The account is bound with user roles and rights. Keep the account information properly and do not disclose the account information to others or exercise corresponding rights on behalf of others
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Six months after the end of the study
Access Criteria: The responsible investigator for the study may be contacted for access to data from this trial
URL: http://www.medresman.org.cn